CLINICAL TRIAL: NCT01337674
Title: A Study to Evaluate the Co-Administration of MK-4618 With Antihypertensive Agents
Brief Title: Co-Administration of MK-4618 With Antihypertensive Agents (MK-4618-010)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4618-010
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide; Metoprolol; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Panel A: MK-4618 + Met → PBO + Met (Experimental): Once daily oral dose of MK-4618 (two 50-mg tablets) on Days 1 through 7 in Period 1 followed by once daily oral dose of placebo (two tablets) on Days 1 through 7 in Period 2. Participants receive previously prescribed daily dose of metoprolol (Met) for the duration of the study. A 2-week washout period follows Period 1.
  Interventions: Drug: MK-4618; Drug: Placebo for MK-4618; Drug: Metoprolol
- Panel A: PBO + Met → MK-4618 + Met (Experimental): Once daily oral dose of placebo (two tablets) on Days 1 through 7 in Period 1 followed by MK-4618 (two 50-mg tablets) on Days 1 through 7 in Period 2. Participants receive previously prescribed daily dose of metoprolol (Met) for the duration of the study. A 2-week washout period follows Period 1.
  Interventions: Drug: MK-4618; Drug: Placebo for MK-4618; Drug: Metoprolol
- Panel B: MK-4618 + Amlo → PBO + Amlo (Experimental): Once daily oral dose of MK-4618 (two 50-mg tablets) on Days 1 through 7 in Period 1 followed by once daily oral dose of placebo (two tablets) on Days 1 through 7 in Period 2. Participants receive previously prescribed daily dose of amlodipine (Amlo) for the duration of the study. A 2-week washout period follows Period 1.
  Interventions: Drug: MK-4618; Drug: Placebo for MK-4618; Drug: Amlodipine
- Panel B: PBO + Amlo → MK-4618 + Amlo (Experimental): Once daily oral dose of placebo (two tablets) on Days 1 through 7 in Period 1 followed by MK-4618 (two 50-mg tablets) on Days 1 through 7 in Period 2. Participants receive previously prescribed daily dose of amlodipine (Amlo) for the duration of the study. A 2-week washout period follows Period 1.
  Interventions: Drug: MK-4618; Drug: Placebo for MK-4618; Drug: Amlodipine

INTERVENTIONS:
Drug: MK-4618 — Once daily oral dose of MK-4618 100 mg (two 50 mg tablets) on Days 1 through 7
Drug: Placebo for MK-4618 — Once daily oral dose of placebo for MK-4618 100 mg (two 50 mg tablets) on Days 1 through 7
Drug: Metoprolol — Previously prescribed daily dose of open-label metoprolol for the duration of the study
  Other Names: Toprol-XL
  Arms: Panel A: MK-4618 + Met → PBO + Met; Panel A: PBO + Met → MK-4618 + Met
Drug: Amlodipine — Previously prescribed daily dose of open-label amlodipine for the duration of the study
  Other Names: Norvasc
  Arms: Panel B: MK-4618 + Amlo → PBO + Amlo; Panel B: PBO + Amlo → MK-4618 + Amlo

SUMMARY:
This study will evaluate the safety and tolerability of MK-4618 when coadministered with antihypertensive agents and will evaluate changes in blood pressure following co-administration of MK-4618 with a beta blocker and a vasodilator. The primary hypothesis of the study is that MK-4618 does not result in a clinically meaningful change in systolic blood pressure relative to placebo when co-administered with a beta-blocker or with amlodipine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female not of childbearing potential
* Not a nursing mother
* Must be on stable dose of a beta blocker (Panel A only) or amlodipine (Panel B only) for the treatment of hypertension for at least 6 weeks prior to enrollment. Must take the designated daily dose of metoprolol or amlodipine for the duration of the study
* In good health other than hypertension
* Nonsmoker
* Participant has a resting systolic blood pressure <150 and >95 mmHg and a diastolic blood pressure <95 and >75 mmHg at prestudy clinical evaluation

Exclusion Criteria:

* Any illness that might confound the results of the study or pose a risk by participation
* History of orthostatic hypotension (decrease in blood pressure upon standing accompanied by symptoms of lightheadedness or dizziness)
* History of cancer, excepting certain skin or cervical cancers or cancers that were treated successfully 10 or more years prior to screening
* Condition for which there is a warning, contraindication, or precaution against the use of extended release metoprolol (Panel A) or amlodipine (Panel B)
* Consumes excessive amounts of alcohol or caffeine daily
* Has multiple and/or severe allergies (including latex allergy) or has had an anaphylactic reaction or significant intolerance to drugs or food
* Uses illicit drugs or has a history of drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2011-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=4618-010&kw=4618-010&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Panel A: MK-4618 + Met → PBO + Met | Panel A: PBO + Met → MK-4618 + Met | Panel B: MK-4618 + Amlo → PBO + Amlo | Panel B: PBO + Amlo → MK-4618 + Amlo
Started | 6 | 7 (The discontinued participant was replaced) | 6 | 7 (The discontinued participant was replaced)
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Discontinued due to blood draws | 0 | 0 | 0 | 1
Period: Two-week Washout Period
Arm/Group | Panel A: MK-4618 + Met → PBO + Met | Panel A: PBO + Met → MK-4618 + Met | Panel B: MK-4618 + Amlo → PBO + Amlo | Panel B: PBO + Amlo → MK-4618 + Amlo
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Panel A: MK-4618 + Met → PBO + Met | Panel A: PBO + Met → MK-4618 + Met | Panel B: MK-4618 + Amlo → PBO + Amlo | Panel B: PBO + Amlo → MK-4618 + Amlo
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panel A Participants: Once daily oral dose of MK-4618 (two 50-mg tablets) or placebo (two tablets) on Days 1 through 7 in Period 1 followed by the crossover treatment in Period 2. Participants receive previously prescribed daily dose of metoprolol for the duration of the study. A 2-week washout period follows Period 1.
- Panel B Participants: Once daily oral dose of MK-4618 (two 50-mg tablets) or placebo (two tablets) on Days 1 through 7 in Period 1 followed by the crossover treatment in Period 2. Participants receive previously prescribed daily dose of amlodipine for the duration of the study. A 2-week washout period follows Period 1.
- Total: Total of all reporting groups
Arm/Group | Panel A Participants | Panel B Participants | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Full Range); unit: Years] | 53.8 [42 to 68] | 55.2 [41 to 77] | 54.5 [41 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Clinical or Laboratory Adverse Experience
Description: An adverse experience was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the sponsor's product is also an adverse experience. The percentage of participants with a clinical or laboratory adverse experience was recorded.
Time Frame: Up to 42 days
Population: The All Subjects as Treated population included all participants who received >=1 dose of study drug
Measure: Number; unit: Percentage of participants
Groups:
- Panel A: MK-4618 + Met: Once daily oral dose of MK-4618 (two 50-mg tablets) in Period 1 or 2. Participants receive previously prescribed daily dose of metoprolol for the duration of the study. A 2-week washout period follows Period 1.
- Panel A: PBO + Met: Once daily oral dose of placebo (two tablets) in Period 1 or 2. Participants receive previously prescribed daily dose of metoprolol for the duration of the study. A 2-week washout period follows Period 1.
- Panel B: MK-4618 + Amlo: Once daily oral dose of MK-4618 (two 50-mg tablets) in Period 1 or 2. Participants receive previously prescribed daily dose of amlodipine for the duration of the study. A 2-week washout period follows Period 1.
- Panel B: PBO + Amlo: Once daily oral dose of placebo (two tablets) in Period 1 or 2. Participants receive previously prescribed daily dose of amlodipine for the duration of the study. A 2-week washout period follows Period 1.
Arm/Group | Panel A: MK-4618 + Met | Panel A: PBO + Met | Panel B: MK-4618 + Amlo | Panel B: PBO + Amlo
Number analyzed (Participants) | 12 | 13 | 12 | 13
Percentage of participants | 33.3 | 53.8 | 41.7 | 61.5

2. Primary Outcome: Maximum Change From Baseline in Semi-recumbent and Standing Systolic Blood Pressure: Panel A
Description: Semi-recumbent and standing systolic blood pressure was measured predose and at intervals up to 24 hours postdose on Day 1 and Day 7. The baseline value is the average of measurements taken in the hour before dosing. Participants were to rest quietly in a semi-recumbent position for at least 10 minutes before each semi-recumbent measurement.
Time Frame: Baseline (predose) and up to 24 hours postdose on Day 1 and Day 7
Population: The All Subjects as Treated population included all participants who received >=1 dose of study drug.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Panel A: MK-4618 + Met | Panel A: PBO + Met
Number analyzed (Participants) | 12 | 13
mmHg
  Semi-recumbent, Day 1 | 16.03 [9.46 to 22.61] | 17.25 [10.93 to 23.57]
  Semi-recumbent, Day 7 | 14.38 [7.81 to 20.96] | 12.10 [5.78 to 18.42]
  Standing, Day 1 | 14.79 [7.43 to 22.15] | 13.14 [6.01 to 20.26]
  Standing, Day 7 | 6.12 [-1.24 to 13.49] | 7.21 [0.09 to 14.34]
Statistical Analysis 1: Comparison: Panel A: MK-4618 + Met vs Panel A: PBO + Met; Semi-recumbent, Day 1; Test type: Non-Inferiority or Equivalence — Hypothesis: the upper bound of the 90% confidence interval for the difference in maximum change from baseline for MK-4618 + Met versus PBO + Met is <20 mmHg; Mean Difference (Final Values) = -1.22, 90% CI 2-sided [-8.42 to 5.98] — The estimated parameter is mean maximum change from baseline for placebo minus MK-4618. Mean and confidence interval for the difference were obtained from linear mixed effects model performed on the maximum increase from baseline values
Statistical Analysis 2: Comparison: Panel A: MK-4618 + Met vs Panel A: PBO + Met; Semi-recumbent, Day 7; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.29, 90% CI 2-sided [-4.92 to 9.49] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Panel A: MK-4618 + Met vs Panel A: PBO + Met; Standing, Day 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.65, 90% CI 2-sided [-5.31 to 8.62] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Panel A: MK-4618 + Met vs Panel A: PBO + Met; Standing, Day 7; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.09, 90% CI 2-sided [-8.06 to 5.88] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Maximum Change From Baseline in Semi-recumbent and Standing Systolic Blood Pressure: Panel B
Description: as for outcome 2
Time Frame: Baseline (predose) and up to 24 hours postdose on Day 1 and Day 7
Population: The All Subjects as Treated population included all participants who received >=1 dose of study drug.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Panel B: MK-4618 + Amlo | Panel B: PBO + Amlo
Number analyzed (Participants) | 12 | 13
mmHg
  Semi-recumbent, Day 1 | 14.69 [9.65 to 19.72] | 12.74 [7.87 to 17.61]
  Semi-recumbent, Day 7 | 10.52 [5.48 to 15.55] | 16.43 [11.56 to 21.30]
  Standing, Day 1 | 6.50 [1.27 to 11.73] | 12.75 [7.70 to 17.79]
  Standing, Day 7 | 6.33 [1.10 to 11.57] | 7.90 [2.85 to 12.95]
Statistical Analysis 1: Comparison: Panel B: MK-4618 + Amlo vs Panel B: PBO + Amlo; Semi-recumbent, Day 1; Test type: Non-Inferiority or Equivalence — Hypothesis: the upper bound of the 90% confidence interval for the difference in maximum change from baseline for MK-4618 + Amlo versus PBO + Amlo is <20 mmHg; Mean Difference (Final Values) = 1.95, 90% CI 2-sided [-2.85 to 6.75] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Panel B: MK-4618 + Amlo vs Panel B: PBO + Amlo; Semi-recumbent, Day 7; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.91, 90% CI 2-sided [-10.71 to -1.11] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Panel B: MK-4618 + Amlo vs Panel B: PBO + Amlo; Standing, Day 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.25, 90% CI 2-sided [-11.47 to -1.03] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Panel B: MK-4618 + Amlo vs Panel B: PBO + Amlo; Standing, Day 7; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.57, 90% CI 2-sided [-6.79 to 3.65] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Steady-state Area Under the Plasma Concentration Versus Time Curve (AUC0-24hr) for MK-4618
Description: Blood samples were collected on Day 7 predose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose for the determination of plasma MK-4618 concentration. The hypothesis for this outcome is that the steady-state AUC0-24hr for MK-4618 is >=0.47 uM*hr.
Time Frame: Predose and up to 24 hours postdose on Day 7
Population: The Per Protocol population included participants who complied with the protocol sufficiently to ensure that the data will likely exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (90% Confidence Interval); unit: uM*hr
Arm/Group | Panel A: MK-4618 + Met | Panel B: MK-4618 + Amlo
Number analyzed (Participants) | 12 | 12
uM*hr | 2.60 [2.09 to 3.24] | 4.60 [3.69 to 5.74]

ADVERSE EVENTS:
Time Frame: Up to 42 days
Arm/Group | Panel A: MK-4618 + Met | Panel A: PBO + Met | Panel B: MK-4618 + Amlo | Panel B: PBO + Amlo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 4/12 | 7/13 | 5/12 | 8/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: MK-4618 + Met (N=12) | Panel A: PBO + Met (N=13) | Panel B: MK-4618 + Amlo (N=12) | Panel B: PBO + Amlo (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 5 (6) | 2 (4) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission